CLINICAL TRIAL: NCT07050940
Title: Anti PD-1 Plus Postbiotic Versus Anti PD-1 Alone in Locally Advanced or Metastatic, Treatment naïve, Cutaneous Melanoma: a Phase II Randomized Study With Correlative Biomarkers' Analysis:
Brief Title: Anti PD-1 Plus Postbiotic Versus Anti PD-1 Alone in Locally Advanced or Metastatic, Treatment naïve, Cutaneous Melanoma Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera di Perugia (Other)
Collaborators: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Mario Mandalà, Director of Department, Azienda Ospedaliera di Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Raffaello-Res
Record Dates: First submitted 2025-03-24; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Melanoma Metastatic
Keywords: melanoma stage IIIC or IV; untreated for metastatic disease
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postbiotic+AntiPD1 (Experimental): patient will be treated with the postbiotic agent and AntiPD1 choose as for standard practice
  Interventions: Dietary Supplement: Postbiotic; Drug: AntiPD1
- AntiPD1 (Active Comparator): patient will be treated with AntiPD1 as per clinical standard practice
  Interventions: Drug: AntiPD1

INTERVENTIONS:
Dietary Supplement: Postbiotic — postbiotic food supplement PostbiotiX-HLA 1 capsule (200mg) /day
  Arms: Postbiotic+AntiPD1
Drug: AntiPD1 — Antibody to PD1 approved for standard of care

SUMMARY:
The association between microbiota and response to ICI-based therapy reflects the ability of bacterial metabolites to upregulate MHC class I APM component expression and/or function in cancer cells, leading to their elimination by the host's immune system.

Thus, the aim of this project is to evaluate the ability of anti PD-1 combined with postbiotic, that here will be a coadjuvant of a standard immunotherapy to upregulate MHC class I APM component expression and/or function in cancer cells compared to anti PD-1 alone in first line advanced melanoma patients.

DETAILED DESCRIPTION:
The study is designed for the primary endpoint as a non-comparative calibrated phase II clinical trial. Patients assigned to the anti PD-1 alone arm will be considered as the calibration group. . Results obtained in the calibration arm will be used to judge the results obtained in the experimental arm.

This is a study protocol settled up on a biological primary endpoint To evaluate the activity of the combination of anti PD-1 plus postbiotic in terms of upregulation of MHC class I APM component expression and/or function in advanced, treatment naïve, cutaneous melanoma patients. The Clinical Objectives is to evaluate the activity of the combination of anti PD-1 plus postbiotic compared to anti PD-1 alone in terms of overall response rate (ORR).

To evaluate the efficacy of the combination of anti PD-1 plus postbiotic compared to anti PD-1 alone in terms of PFS.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Histologically confirmed, unresectable stage IIIC or IV metastatic melanoma;
* Eastern Cooperative Oncology Group performance status of 0 or 1;
* The patient must treatment naïve for metastatic disease
* Patients who have received anti-PD-1 therapy or anti BRAF/MEK in adjuvant setting and relapsed after 6 months of ending adjuvant therapy are allowed to enter clinical study.
* Patient has at least one measurable lesion that qualifies as a target lesion based on RECIST 1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
* Patient is willing to undergo a pretreatment tumor biopsy or provide qualifying archival tumor tissue. To qualify, archival tissue must have been sampled after last exposure to any systemic anti-neoplastic agent (including TVEC or anti-PD-L1 therapy whichever is last). Patients unable to undergo a biopsy may be enrolled if risk/benefit ratio of biopsy is considered unfavorable and/or when a biopsy would likely lead to significant delays in care. This decision must be accompanied by supporting documentation from the Investigator and performed in consultation with Medical Monitor. All pretreatment tissue must have been collected no more than 120 days prior to screening.
* Patient has recovered from the effects of any previous chemotherapy, immunotherapy, other prior systemic anticancer therapy, radiotherapy, and/or surgery (ie, residual toxicity no worse than Grade 1 [Grade 2 treatment-associated peripheral neuropathy and/or any grade of alopecia are acceptable assuming all other inclusion criteria are met]).
* Patient who has received prior systemic anti-neoplastic agent(s) must wait at least 5 half-lives or 4 weeks (whichever is shorter) following prior therapy before enrollment into the study, or 4 weeks if the half-life of a given investigational agent is not known.
* Patient has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 within 5 days before the first dose of study drug and an estimated life expectancy of at least 3 months.
* Patient has adequate hematologic reserve as evidenced by:

Absolute neutrophil count (ANC) of ≥1000/μL, Absolute lymphocyte count of

≥500/μL, Platelet count of ≥75,000/μL, and Hemoglobin of ≥9 g/dL (patients may be transfused to this level, if necessary, but transfusion must occur >1 week prior to the first dose of study drug).

* Patient has adequate hepatic function as evidenced by aspartate transaminase and alanine transaminase values ≤3 × the upper limit of normal (ULN) and serum total bilirubin values of ≤1.5 × ULN (≤2 × ULN for patients with known Gilbert's syndrome) for the reference laboratory measured within 7 days prior to the first dose of study drug. For patients with documented baseline liver metastasis, the following limits will apply: 5 × ULN for transaminase and 2 × ULN for bilirubin.
* Patient has adequate renal function as evidenced by a serum creatinine ≤1.5 × the ULN for the reference laboratory or a calculated creatinine clearance of ≥45 mL/min by the Cockcroft-Gault Equation measured within 7 days prior to the first dose of study drug.
* Patient has international normalized ratio (INR) AND/OR prothrombin time (PT) AND activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless the patient is receiving anticoagulant therapy, in which case INR and/or PT and aPTT must be within the desired therapeutic range of intended use for such anticoagulants.
* Patient agrees to abide by the contraceptive requirements detailed in the protocol.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test (serum or urine) within 3 days before the first dose of study drug (see the protocol for the definition of WOCBP).
* Life expectancy more than 3 months
* Presence of instrumentally or clinically measurable or evaluable lesions Informed consent obtained

Exclusion Criteria:

* Patients with mucosal or with a primary ocular melanoma
* Active symptomatic or asymptomatic brain metastases
* Patients with the following disorders: active, known, or suspected autoimmune disease (except for some non-serious disorders, such as vitiligo and type 1 diabetes mellitus, as specified in the study protocol);
* Previous malignancies (exceptions skin basocellular or squamocellular carcinoma radically resected, in situ uterine cervix in situ carcinoma radically resected) in the previous 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Biological response rate | 18 months
  proportion of responder patients at 12 weeks from treatment start. The response to treatment is based on the IHC level of HLA and NRLC5 at baseline and after 12 weeks from treatment start. An IHC level equal to 0 or 1+ is defined as low, while a IHC value equal to 2+ or 3+ is defined as high

SECONDARY OUTCOMES:
Objective Response Rate | 18 months
  the proportion of patients with a complete (CR) or partial response (PR) as best response during treatment as determined by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Mandalà, MD, Principal Investigator — AO perugia-University of perugia
Locations (5):
- Italy (5):
  - Bari University-Oncologia medica, Bari, BA
  - Torino University-Le Molinette, Torino, TO
  - IRCCS Papa Giovanni II Bari, Bari
  - INT Milano, Milan
  - AO Perugia, Perugia

IPD SHARING:
Plan to Share IPD: No
only for patient referral to italian site

REFERENCES:
- [Background] Ferrari V, Lo Cascio A, Melacarne A, Tanaskovic N, Mozzarelli AM, Tiraboschi L, Lizier M, Salvi M, Braga D, Algieri F, Penna G, Rescigno M. Sensitizing cancer cells to immune checkpoint inhibitors by microbiota-mediated upregulation of HLA class I. Cancer Cell. 2023 Oct 9;41(10):1717-1730.e4. doi: 10.1016/j.ccell.2023.08.014. Epub 2023 Sep 21. PMID 37738976